CLINICAL TRIAL: NCT03597750
Title: Pressure Ulcer Prevention Using Static Air Support Devices (Repose®) Versus Alternating-Pressure Devices in a High Risk Population in Nursing Homes: A Multi-Center Prospective Randomized Controlled Trial and Qualitative Study
Brief Title: Comparison of Static Air Support Devices (Repose®) and Alternating-Pressure Devices in the Prevention of Pressure Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Frontier Medical Group, UK (Unknown)
Responsible Party: Principal Investigator, UCVV, University Centre for Nursing and Midwifery, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EC/2017/0266; B670201731706 (Other: Ethics Committee UZ Gent)
Record Dates: First submitted 2017-10-23; First posted 2018-07-24 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Pressure Ulcer; Pressure Injury; Pressure Sore; Bed Sore
Keywords: Static air support devices; Alternating-pressure devices; High risk population; Elderly; Prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static air support devices (Repose®) (Experimental): Alternating-pressure devices will be replaced by static air support devices (Repose®) during 14 days:
  * Repose® Mattress
  * Repose® Cushion
  * Repose® Wedge or Foot Protectors
  The frequency of repositioning remains unchanged.
  Interventions: Device: Repose®
- Alternating-pressure devices (No Intervention): Instead of replacing the alternating-pressure devices by static air support devices (Repose®), the residents remain on their alternating-pressure devices.
  The frequency of repositioning remains unchanged.

INTERVENTIONS:
Device: Repose® — * Repose® Mattress
  * Repose® Cushion
  * Repose® Wedge or Foot Protectors
  Arms: Static air support devices (Repose®)

SUMMARY:
Maintaining and improving skin health are major goals in acute and long-term care. Patients at the extremes of age, the critically ill, medically compromised and those with immobility are at risk for developing several skin disorders, with pressure ulcers (PUs) as one of the most common and mostly preventable ones. Prevalence figures of PUs vary between 6.4% and 31.4%. PUs are described as localised injuries to the skin and/or underlying tissue, usually over a bony prominence, as a result of pressure or pressure combined with shear. Prevention of PUs is internationally seen to be a key quality indicator of care. To prevent PUs, reducing both the amount and the duration of pressure and shear at the pressure points of the body is strongly recommended. One of the interventions to achieving this, is the use of pressure-reducing devices (mattresses, cushions, etc.). Studies that compare the (cost-) effectiveness of different pressure-reducing devices are needed.

The primary aim of this study is to compare the (cost-) effectiveness of pressure ulcer prevention in high risk patients using static air support devices (Repose®) versus alternating-pressure devices. The second aim is to get insight in patients' experiences and perceptions of comfort using static air support devices and alternating-pressure devices. The third aim is to get insight in caretakers' perceptions of barriers and facilitators of the use of static air support devices and alternating-pressure devices and to reveal how these perceptions influence the readiness to use the products in clinical practice.

This randomized controlled trial will be performed in ca. 25 nursing homes in a random sample of 306 residents who are at high risk of developing pressure ulcers. Residents will be included in the study for a period of 14 days. Skin assessment and risk factor registration will be done on a daily basis by the nurses. Reliability checks and time measurements will be completed by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* High risk of pressure ulcers (Braden score < 12) and/or pressure ulcer category 1
* Currently using alternating-pressure devices
* Bedbound (> 8 hours in bed) or chair bound (> 8 hours in chair)
* Aged > 65 years

Exclusion Criteria:

* Pressure ulcer category 2,3,4, deep tissue injury (DTI) or unstageable pressure ulcer
* Expected length of stay < 2 weeks
* End of life care
* Medical contraindication for use of static air support devices

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 308 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence (Cat. II+) | 14 days
  Development of at least 1 pressure ulcer Cat. II+ during study period

SECONDARY OUTCOMES:
Patient experiences and perceptions using a static air mattress | 14 days
  Patients experiences and perceptions of comfort using static air support devices and alternating-pressure mattresses. Patient acceptability [tolerance, (sleep) comfort, pain)
Caretakers perceptions of barriers and facilitators to use static air mattress | 14 days
  Nurses acceptability [barriers and facilitators].
Incidence of incontinence-associated dermatitis (IAD) | 14 days
  Development of at least 1 IAD during study period
Cost of the intervention (Repose) versus the standard care (Alternating) | 14 days
  Economic measures (from an organizational and patient perspective)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, PhD, Principal Investigator — University Ghent
Locations (26):
- Belgium (26):
  - Woonzorgcentrum Zonnetij, Aartselaar, Antwerpen
  - Woonzorgcentrum Zonnewende, Aartselaar, Antwerpen
  - Woonzorgcentrum De Mick, Brasschaat, Antwerpen
  - Woonzorgcentrum Sint-Maria, Brecht, Antwerpen
  - Woonzorgcentrum Veilige Have, Aalter, Oost-Vlaanderen
  - Woonzorgcentrum Sint-Jozef, Assenede, Oost-Vlaanderen
  - Woonzorgcentrum De Vijvers, Gentbrugge, Oost-Vlaanderen
  - Woonzorgcentrum Meulenbroek, Hamme, Oost-Vlaanderen
  - Woonzorgcentrum Heilig Hart, Oudenaarde, Oost-Vlaanderen
  - Woonzorgcentrum Egmont, Zottegem, Oost-Vlaanderen
  - Woonzorgcentrum Sint-Vincentius, Avelgem, West-Vlaanderen
  - Woonzorgcentrum Hallenhuis, Bruges, West-Vlaanderen
  - Woonzorgcentrum Minnewater, Bruges, West-Vlaanderen
  - Woonzorgcentrum Ter Potterie, Bruges, West-Vlaanderen
  - Woonzorgcentrum Van Zuylen, Bruges, West-Vlaanderen
  - Woonzorgcentrum Huize Zonnelied, Ieper, West-Vlaanderen
  - Woonzorgcentrum Maria Rustoord, Ingelmunster, West-Vlaanderen
  - Woonzorgcentrum De Plataan, Izegem, West-Vlaanderen
  - Woonzorgcentrum De Pottelberg, Kortrijk, West-Vlaanderen
  - Woonzorgcentrum Sint-Jozef, Kortrijk, West-Vlaanderen
  - Woonzorgcentrum OLV Gasthuis, Poperinge, West-Vlaanderen
  - Woonzorgcentrum Hof Ten Ijzer, Reninge, West-Vlaanderen
  - Woonzorgcentrum Wintershove, Vlamertinge, West-Vlaanderen
  - Woonzorgcentrum De Meers, Waregem, West-Vlaanderen
  - Woonzorgcentrum Sint-Camillus, Wevelgem, West-Vlaanderen
  - Woonzorgcentrum Sint-Amand, Zwevegem, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McInnes E, Jammali-Blasi A, Bell-Syer SE, Dumville JC, Middleton V, Cullum N. Support surfaces for pressure ulcer prevention. Cochrane Database Syst Rev. 2015 Sep 3;2015(9):CD001735. doi: 10.1002/14651858.CD001735.pub5. PMID 26333288
- [Background] Serraes B, Beeckman D. Static Air Support Surfaces to Prevent Pressure Injuries: A Multicenter Cohort Study in Belgian Nursing Homes. J Wound Ostomy Continence Nurs. 2016 Jul-Aug;43(4):375-8. doi: 10.1097/WON.0000000000000244. PMID 27391289
- See also: Website of the research group — http://www.ucvvgent.be